CLINICAL TRIAL: NCT06984939
Title: Use of a Handheld Tool for Active Distraction of Children and Adolescents During Painful Procedures
Brief Title: A Handheld Tool for Active Distraction of Children and Adolescents During Painful Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Principal Investigator, Mette Engan, Principal Investigator, Haukeland University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 873256
Record Dates: First submitted 2025-05-20; First posted 2025-05-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pain
Keywords: Active distraction; Procedural pain; Pediatrics
MeSH Terms: conditions — Pain; Pain, Procedural | interventions — Hand Strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Grasp (Experimental): Participants assigned to the Grasp arm will be instructed to use Grasp during the procedure.
  Interventions: Device: Grasp

INTERVENTIONS:
Device: Grasp — Participants assigned to the intervention group will be instructed to squeeze the Grasp ball at regular intervals of approximately every 1-2 seconds. This action will activate a melody played through a speaker connected to the iPad, accompanied by a dynamic wavy line displayed on the screen. Participants will begin squeezing the Grasp ball at least 10 seconds prior to the start of the procedure and will continue until the procedure is completed.
  Other Names: Active distraction
  Arms: Grasp

SUMMARY:
The goal of this clinical trial is to learn if the handheld device Grasp, works to reduce pain and distress during small procedures involving a needle prick in children and adolescents. The main question it aims to answer is:

Does repetitive squeezing of the Grasp device during the painful procedure affect self-reported pain and distress?

Researchers will compare using the Grasp device during procedures where children and adolescent are having a needle prick (venous puncture, insertion of a peripheral venous catheter, local anesthetic injection before dental treatment) with standard care, to see if Grasp works to reduce pain and distress.

Participants will:

* Use Grasp or standard care during procedures involving a needle prick
* Report pain and distress on a paper form before and after the procedure

DETAILED DESCRIPTION:
This project seeks to contribute to the evidence base regarding the utility of active distraction techniques, such as Grasp, in pediatric clinical settings. Findings may inform the development of non-pharmacological interventions aimed at improving the patient experience and reducing procedural distress among children.

Grasp is a communication tool comprising both hardware and software components. The hardware consists of a handheld, soft silicone ball embedded with pressure sensors capable of detecting squeezes of varying intensity and duration. The software component is a dedicated application designed for use on an iPad, which forms an integral part of the system. Squeezing the ball generates visual and auditory feedback in real time via the application, presented through dynamic curves and sound cues, including musical elements. Data from the pressure sensors is transmitted live to the software via Bluetooth, enabling immediate sensory feedback. Grasp is CE-marked and registered as a medical device under ID NO918873724/0943-55311 by the Norwegian Directorate of Medical Products.

The primary objective of this study is to evaluate the efficacy of Grasp as an active distraction tool in reducing perceived pain and distress in children undergoing minor but potentially distressing medical procedures. We aim to recruit children aged 8-15 years from Children and Youth Clinic (CYC) at Helse Bergen HF, Helsebanken General Practice, and TkVestland Dental Center. The procedures involved include peripheral venous cannulation (CYC), venipuncture for blood sampling (Helsebanken), and administration of local anesthesia via injection (dental clinic). Participants will be allocated using block randomization. The intervention group will engage with the Grasp system by repeatedly squeezing the ball before and during the procedure, triggering musical feedback. The control group will undergo standard care without the use of Grasp.

We aim to recruit 50 participants at CYC, 50 participants at TK Vestland dental clinic and 20 participants at Helsebanken General Practices.In addition, we will explore the use of Grasp in six patients admitted to hospital with a newly diagnosed diabetes mellitus type 1 who will use Grasp during blood sugar measurement or subcutaneous insulin administration. (These six participants will not participate in the randomized controlled part of the study.)

The primary outcome measure will be self-reported pain, assessed using a combined visual analogue scale (VAS) and numeric rating scale (NRS) (0-10). The secondary outcomes will include self-reported distress, measured using a combined VAS/NRS scale, as well as parents' or legal guardians' assessments of their child's pain and distress, also rated on a similar scale. Additionally, six participants recruited at CYC who have prior experience with peripheral venous cannulation and underwent the procedure using Grap, will be invited to take part in individual semi-structured interviews. These interviews will explore their subjective experiences with the intervention.

The participant will fill out a paper form questionnaire prior to randomization regarding their prior experience, anticipated pain and how anxious they are about the upcoming procedure. Immediately after the needle prick procedure participants and parents will fill out the second form regarding their experience during this procedure. The participant at the dental office will be offered to use the Grasp further through the dental treatment and all participants and parents at the dental office will complete a final similar questionnaire after the completion of dental treatment.

Multiple linear regression analyses will performed to examine the impact of the intervention adjusted for baseline scores. Statistical analyses will be done in R version 4.2.3. Systematic text condensation will be used to analyse the interviews.

ELIGIBILITY:
Inclusion Criteria:

* Written consent has been obtained from the parents or legal guardians.
* Age 8-15 years old

One of the following:

1. Attend the Child and Youth Clinic at Haukeland University Hospital for peripheral venous cannula insertion
2. Attend the Helsebanken in Øystese for blood sampling
3. Attend TKVestland for planned dental treatment involving local anesthesia administered via injection (needle)
4. Admitted to the Child and Youth Clinic at Haukeland University Hospital for the first time due to type 1 diabetes mellitus, requiring frequent blood glucose measurements and insulin injections.

Exclusion Criteria:

* Moderate to severe intellectual disability
* Impaired vision or hearing
* Does not understand the Norwegian language
* General condition affected by illness
* Anticipated use of sedation during the procedure (e.g., Midazolam)
* Previous participation in this study

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported pain | Immediately after the procedure has been completed.
  Self-reported by a combined visual analogue scale and numerical rating scale (0-10)

SECONDARY OUTCOMES:
Self-reported distress | Reported immediately after the procedure has been completed
  Self-reported by a combined visual analogue scale and numeric rating scale ( 0-10)
Parental-reported pain and distress | Reported immediately after the procedure has been completed
  Reported by a combined visual analogue scale and numeric rating scale ( 0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Mette Engan, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inan G, Inal S. The Impact of 3 Different Distraction Techniques on the Pain and Anxiety Levels of Children During Venipuncture: A Clinical Trial. Clin J Pain. 2019 Feb;35(2):140-147. doi: 10.1097/AJP.0000000000000666. PMID 30362982
- [Background] McGrath PJ, Walco GA, Turk DC, Dworkin RH, Brown MT, Davidson K, Eccleston C, Finley GA, Goldschneider K, Haverkos L, Hertz SH, Ljungman G, Palermo T, Rappaport BA, Rhodes T, Schechter N, Scott J, Sethna N, Svensson OK, Stinson J, von Baeyer CL, Walker L, Weisman S, White RE, Zajicek A, Zeltzer L; PedIMMPACT. Core outcome domains and measures for pediatric acute and chronic/recurrent pain clinical trials: PedIMMPACT recommendations. J Pain. 2008 Sep;9(9):771-83. doi: 10.1016/j.jpain.2008.04.007. Epub 2008 Jun 17. PMID 18562251
- [Background] Birnie KA, Noel M, Chambers CT, Uman LS, Parker JA. Psychological interventions for needle-related procedural pain and distress in children and adolescents. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005179. doi: 10.1002/14651858.CD005179.pub4. PMID 30284240
- [Background] Shen T, Wang X, Xue Q, Chen D. Active versus passive distraction for reducing procedural pain and anxiety in children: a meta-analysis and systematic review. Ital J Pediatr. 2023 Aug 31;49(1):109. doi: 10.1186/s13052-023-01518-4. PMID 37653423
- See also: Information about the study — https://www.helse-bergen.no/kliniske-studier/bruk-av-et-handholdt-verktoy-for-aktiv-avledning-av-barn-og-unge-ved-ubehagelige-prosedyrer/